CLINICAL TRIAL: NCT06501287
Title: Postprandial Triglyceride Impact on Coronary Atherosclerosis in Non-Diabetic Patient in Sohag University Hospital [NCT ID Not Yet Assigned]
Brief Title: Postprandial Triglyceride Impact on Coronary Atherosclerosis in Non-Diabetic Patient in Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Fatma Madhy Eissa (Other)
Responsible Party: Sponsor-Investigator, Fatma Madhy Eissa, resident internal medecine, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh-Med-24-04-02Ms
Record Dates: First submitted 2024-05-20; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Coronary Atheroscleroses
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group I (control group):: patients with normal coronary angiography and normal postprandial triglycerides
  Interventions: Diagnostic Test: Postprandial triglyceride
- Group II: : patients with abnormal coronary angiography and high level of postprandial triglycerides more than 200mg/dl. They will be divided into subgroups according to severity of coronary artery disease (mild, moderate and severe) according to (Syntax score)
  Interventions: Diagnostic Test: Postprandial triglyceride
- Group III: : patients with abnormal coronary angiography and normal postprandial triglycerides.
  Interventions: Diagnostic Test: Postprandial triglyceride

INTERVENTIONS:
Diagnostic Test: Postprandial triglyceride — impact of postprandial triglyceride level on coronary atherosclerosis

SUMMARY:
INTRODUCTION Cardiovascular diseases, including coronary artery disease (CAD), are the leading cause of mortality worldwide. Despite remarkable advancements in diagnostic and therapeutic approaches, CAD continues to pose formidable challenges. Atherosclerosis, characterized by the deposition of lipids, inflammatory cells, and fibrous tissue within the arterial walls, is the fundamental pathology underpinning CAD. Atherosclerosis development and progression are closely intertwined with lipid metabolism, particularly elevated levels of low-density lipoprotein cholesterol (LDL-C) and reduced levels of high-density lipoprotein cholesterol (HDL-C) *1+. However, emerging evidence suggests that postprandial triglyceride levels, the transient increase in triglycerides following a meal, may play a pivotal role in atherosclerotic processes *2+. Postprandial hypertriglyceridemia has been linked to various cardiovascular risk factors, including inflammation, endothelial dysfunction, oxidative stress, and altered hemostasis *3+. cardiovascular disease (CVD) causes death for 4 million subjects in Europe every year. It causes death for women *2.2 million (55%)+ than men *1.8 million (45%)+, and cardiovascular (CV) deaths under 65 years more prevalent in men (490 000 versus 193 000) *4+. Endothelial dysfunction was the main cause of vascular atherosclerosis. The damage of Endothelium cause lipids and macrophages accumulation (mostly lowdensity lipoprotein) in vessel injury site *5+. Lipids considered the major cause of atherosclerosis *6+. The increase of blood cholesterol (especially LDL) considered the main cause of the disease. High levels of triglycerides could be independent risk factor for coronary artery disease (CAD), particularly in women. Although, it was suggested that high level of density lipoproteins (HDLs) can prohibit these risk factors. Extensive examinations showed that lipid decrease the prevention of CAD in primary and secondary cases *7+. The level > 90% of total glyceride and/or LDL and level > 10% of HDL confirm dyslipidemia *8+

ELIGIBILITY:
Inclusion criteria includes CAD based on coronary angiography, laboratory and ECG evidence.

Exclusion criteria:

Patients with other co-morbidities diseases, such as liver and kidney disorders and thyroid diseases. Diabetic patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: includes CAD based on coronary angiography, laboratory and ECG evidence.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
impact of postprandial triglyceride level on coronary atherosclerosis in non diabetic patients | 7 months
  impact of postprandial triglyceride concentration measured by chemistry analyzer on coronary atherosclerosis (assassed by plaque volume and luminal narrowing in coronary angiography )in non-diabetic patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Background] Nordestgaard BG, Benn M, Schnohr P, Tybjaerg-Hansen A. Nonfasting triglycerides and risk of myocardial infarction, ischemic heart disease, and death in men and women. JAMA. 2007 Jul 18;298(3):299-308. doi: 10.1001/jama.298.3.299. PMID 17635890
- [Background] Tushuizen ME, Nieuwland R, Scheffer PG, Sturk A, Heine RJ, Diamant M. Two consecutive high-fat meals affect endothelial-dependent vasodilation, oxidative stress and cellular microparticles in healthy men. J Thromb Haemost. 2006 May;4(5):1003-10. doi: 10.1111/j.1538-7836.2006.01914.x. PMID 16689751
- [Background] Catapano AL, Graham I, De Backer G, Wiklund O, Chapman MJ, Drexel H, Hoes AW, Jennings CS, Landmesser U, Pedersen TR, Reiner Z, Riccardi G, Taskinen MR, Tokgozoglu L, Verschuren WMM, Vlachopoulos C, Wood DA, Zamorano JL, Cooney MT; ESC Scientific Document Group. 2016 ESC/EAS Guidelines for the Management of Dyslipidaemias. Eur Heart J. 2016 Oct 14;37(39):2999-3058. doi: 10.1093/eurheartj/ehw272. Epub 2016 Aug 27. No abstract available. PMID 27567407